CLINICAL TRIAL: NCT03475927
Title: Knowledge and Awareness of Radiation Hazard in Health-care Personnel; A Quaternary-care Academic Center Study
Brief Title: Knowledge and Awareness of Radiation Hazard in Health-care Personnel
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaowanan Khamtuikrua, Principal Investigator, Mahidol University
Other Study IDs: SI2018-03
Record Dates: First submitted 2017-12-31; First posted 2018-03-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Radiation Hazard

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Concerning and knowledge about radiation hazard questionnaire — Concerning and knowledge about radiation hazard questionnaire to determine the concerning and knowledge of radiation hazard among surgeon and anesthesiologist

SUMMARY:
Knowledge and awareness of radiation hazard in health-care personnel; A Quaternary-care academic center study Aim: To determine knowledge and concerning about radiation hazard in anesthetic personnel and surgeon

study decide: questionnaire based study to ask concerning and knowledge about radiation hazard

ELIGIBILITY:
Inclusion Criteria:

* Anesthetic personnel
* Surgeon: urology, orthopedic, cardiothoracic, neurosurgeon, general

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: anesthetic personnel and surgeon who contact riadiation equipment
Sampling Method: Non-Probability Sample
Enrollment: 214 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
score of multiple choice question test about radiation hazard knowledge in anesthetic personnel and surgeon | 1 year
  score of MCQ test, good knowledge will be determine if more than 9 point of 15 point

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Siriraj hospital, Bangkok, Thailand